CLINICAL TRIAL: NCT00740935
Title: Impact of Systematic Infants Vaccination Against Rotavirus on Gastroenteritis Hospitalization: a Prospective Study in Brest District, France.
Acronym: IVANHOE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: MCM Vaccines B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RB 06.117
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2012-06

CONDITIONS: Rotavirus Gastroenteritis
Keywords: prevention; rotavirus vaccine; gastroenteritis; systematic vaccination; infants; aged 6 to 12 weeks
MeSH Terms: conditions — Gastroenteritis | interventions — RotaTeq

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Cohort of vaccinated infants against rotavirus
  Interventions: Biological: Rotateq vaccine

INTERVENTIONS:
Biological: Rotateq vaccine — Vaccination against rotavirus
  Three oral doses (2 mL) between 6 to 26 weeks of life with at least 4 weeks between each dose.
  Other Names: Rotateq

SUMMARY:
Universal rotavirus vaccination program for infants born in Brest after February 2007, applied by the Centers for Maternal and Infant Health Protection, pediatricians and general practitioners.

Prospective surveillance of hospitalizations for gastroenteritis within the Pediatric Units of Brest University Hospital with systematic testing for Rotavirus.

Evaluation of the impact of the vaccination program on rotaviral gastroenteritis hospitalizations from 2007-2008 and 2008-2009, by comparison with epidemiological data from 2002-2007 in the absence of vaccination.

The principal judgement criterion is the number of pediatric hospitalizations for rotaviral GEA during the 2008-2009 epidemic in children A) under the age of 2 and B) residing in the suburbs of Brest.

ELIGIBILITY:
Inclusion Criteria:

* infants aged 6 to 12 weeks
* born in Brest District, France
* born between Feb 01, 2007 and Nov 19, 2009

Exclusion Criteria:

* contraindication to rotavirus vaccine

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7204 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Hospitalization for gastroenteritis | 2 years

SECONDARY OUTCOMES:
Emergency department consultation for gastroenteritis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud GAGNEUR, Doctor, Study Director — University Hospital, Brest
Locations (1):
- Clinical Investigation Center, Brest, France

REFERENCES:
- [Derived] Roue JM, Nowak E, Le Gal G, Lemaitre T, Oger E, Poulhazan E, Giroux JD, Garenne A, Gagneur A. Impact of rotavirus vaccine on premature infants. Clin Vaccine Immunol. 2014 Oct;21(10):1404-9. doi: 10.1128/CVI.00265-14. Epub 2014 Jul 30. PMID 25080553
- [Derived] Gagneur A, Nowak E, Lemaitre T, Segura JF, Delaperriere N, Abalea L, Poulhazan E, Jossens A, Auzanneau L, Tran A, Payan C, Jay N, de Parscau L, Oger E; IVANHOE investigators. Impact of rotavirus vaccination on hospitalizations for rotavirus diarrhea: the IVANHOE study. Vaccine. 2011 May 12;29(21):3753-9. doi: 10.1016/j.vaccine.2011.03.035. Epub 2011 Apr 13. PMID 21443962